CLINICAL TRIAL: NCT01336582
Title: Phase I Trial to Compare Pharmacokinetics and Safety of SYP-0704A With Taxotere in Subjects With Advanced Solid Tumor
Brief Title: Pharmacokinetic Study of SYP-0704A and Taxotere to Treat Patient With Advanced Solid Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DOCXN101
Record Dates: First submitted 2011-03-21; First posted 2011-04-18 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Solid Tumor
Keywords: suitable candidate; single agent docetaxel therapy; Advanced Solid Tumor
MeSH Terms: interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- docetaxel (Experimental)
  Interventions: Drug: taxotere
- Taxotere (Active Comparator): Docetaxel-PM 75 mg/m2 (70 mg/m2 for age of ≥ 65) Taxotere 75mg/m2 (70 mg/m2 for age of ≥ 65)
  Interventions: Drug: taxotere

INTERVENTIONS:
Drug: taxotere — 70 mg/m2 for age of ≥ 65

SUMMARY:
Primary Objective: Evaluation of the pharmacokinetic equivalence of two Docetaxel formulations in terms of AUC and Cmax.

DETAILED DESCRIPTION:
Comparison of pharmacokinetic parameters (T1/2β, CL, Vdss) Safety as measured by adverse events

ELIGIBILITY:
Inclusion Criteria:

* Subjects who aged 18 years or older.
* Subjects whose written informed consent was obtained complying with the local regulatory requirements prior to their participation in the trial.
* Subjects who have histologically or cytologically confirmed advanced solid tumor.
* Subjects who are a suitable candidate for single agent docetaxel therapy for their advanced solid tumors that have failed to standard therapy.
* Subjects who have fully recovered from reversible toxic effects of prior therapy. The prior chemotherapy, immunotherapy, hormone therapy, surgery, and/or radiotherapy should be completed at least 21 days before the first administration of investigational product.

Exclusion Criteria:

* Subjects who have had a major surgery other than tumor ablation within 2 weeks prior to the screening/baseline visit.
* Subjects who have a history of metastasis or currently have a metastasis to the central nervous system (CNS).
* Subjects who have a preexisting sensory or motor neuropathy of grade ≥ 2 based on NCI CTCAE V3.0.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-08; Primary Completion 2012-04 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of SYP-0704A and Taxotere in terms of AUC | 3 months

SECONDARY OUTCOMES:
Pharmacokinetics of the T1/2 of SYP-0704A and Taxotere | 3 months
Pharmacokinetics of the CL of SYP-0704A and Taxotere | 3 months
Pharmacokinetics of the Vdss of SYP-0704A and Taxotere | 3 months
Number of paticipants with Adverse Events | 3months

CONTACTS AND LOCATIONS:
Overall Officials: Shin je gook, doctor, Principal Investigator — Inje Pusan Paik university hospital
Locations (1):
- Inje Pusan paik University hospital, Pusan, Jin-Gu, South Korea